CLINICAL TRIAL: NCT01216787
Title: A Pilot Trial to Evaluate the Molecular Effects of RO4929097 as Neoadjuvant Therapy for Resectable Stage IIIB, IIIC or IV Melanoma
Brief Title: RO4929097 in Treating Patients With Stage IIIB, Stage IIIC, or Stage IV Melanoma That Can Be Removed by Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study drug not available.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02512; 10-01704; N01CM62204 (NIH); CDR0000685418 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Stage IIIB Melanoma; Stage IIIC Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (gamma-secretase inhibitor RO4929097, surgery) (Experimental): Patients receive oral RO4929097 once daily on days 1-3, 8-10, and 15-17. Within 35-56 days after completion of therapy, patients with stable or responsive disease undergo surgery. Patients may continue RO4929097 for 28 days after surgery in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Other: pharmacological study; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097
  Other Names: R4733; RO4929097
Other: pharmacological study
  Other Names: pharmacological studies
Procedure: therapeutic conventional surgery
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot phase II trial is studying how well RO4929097 works in treating patients with stage III, or stage IV melanoma that can be removed by surgery. RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the molecular effects of Notch signaling inhibition using gamma-secretase inhibitor RO4929097 (RO4929097) in patients with resectable stage IIIB, IIIC, or IV intact melanoma tumors in the neoadjuvant setting.

SECONDARY OBJECTIVES:

I. Assess any indication of clinical activity of RO4929097 in these patients. II. Assess the effect of RO4929097 on Akt-mediated downstream biomarkers in melanoma tissue.

III. Assess the effect of RO4929097 on the melanoma stem cell subpopulation. IV. Identify patient-specific micro-RNA signatures that may correlate with response to therapy, recurrence, and overall survival.

V. Determine the clinical feasibility of measuring circulating melanoma tumor cells in the blood and correlating levels with recurrence and/or survival.

VI. Correlate the shedding of collagen cryptic epitopes in the serum and urine with tumor response and risk of recurrence.

VII. Measure the pharmacokinetics and pharmacodynamics of RO4929097 in these patients.

VIII. Evaluate the impact of RO4929097 on serum markers of angiogenesis. IX. Measure serum autoimmune biomarkers and correlate with clinical response and outcome in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral gamma-secretase inhibitor RO4929097 (RO4929097) once daily on days 1-3, 8-10, and 15-17. Within 35-56 days after completion of therapy, patients with stable or responsive disease undergo surgery. Patients may continue RO4929097 for 28 days after surgery in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor tissue biopsies at baseline and after completion of study therapy for 4E-BP1 and Akt-mediated downstream biomarkers, stem cell subpopulation, and patient-specific micro-RNA signatures studies by IHC and PCR assays. Blood and urine samples are also collected at baseline and periodically during study for pharmacokinetic and pharmacodynamic studies, circulating melanoma endothelial cells and progenitor cell levels, collagen cryptic epitopes, serum markers of angiogenesis, and autoimmune biomarker analysis by ELISA.

After completion of study therapy, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed melanoma

  * Stage IIIB, IIIC, or IV disease
  * Disease that is deemed resectable by surgical consultation

    * Patients must agree to pretreatment biopsies of their tumor
* Measurable disease defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20 mm by conventional techniques OR as ≥ 10 mm by spiral CT scan

  * Measurable lesions must be deemed resectable
  * Skin metastases must be photographed and measured
  * No non-target disease
* No known brain metastases
* Life expectancy > 3 months
* ECOG performance status 0-2 (Karnofsky 60-100%)
* WBC ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 75,000/mm³
* Hemoglobin > 10 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Fertile patients must agree to use 2 forms of contraception (i.e., barrier contraception and 1 other method of contraception) for ≥ 4 weeks prior to, during, and for ≥ 12 months post-treatment
* Negative pregnancy test
* Not pregnant or nursing
* No history of allergic reactions attributed to compounds of similar chemical or biological composition of gamma-secretase inhibitor RO4929097 or other agents used in the study
* No malabsorption syndrome or other condition that would interfere with intestinal absorption
* Able to swallow tablets
* No known history of hepatitis or have a history of liver disease or other forms of cirrhosis
* No uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia, or hypokalemia despite adequate electrolyte supplementation
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia other than chronic
  * Unstable atrial fibrillation
  * Psychiatric illness and/or social situations that would limit compliance with study requirements
* No baseline QTcF > 450 msec (male) or QTcF > 470 msec (female)
* No history of cancer within the past 5 years except curatively treated basal or squamous cell cancer of the skin, in situ cervical cancer, or lobular carcinoma in situ of the breast
* No other concurrent anticancer agents or therapies
* More than 4 weeks since prior immunotherapy or local radiotherapy and recovered
* No prior chemotherapy for melanoma
* No concurrent medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®)
* No concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent ketoconazole or grapefruit juice while taking gamma-secretase inhibitor RO4929097
* No concurrent granulocyte colony-stimulating factors
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Molecular effects of notch-signaling inhibition | Up to 2 years
  All statistics will be descriptive.

SECONDARY OUTCOMES:
Toxicity as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 2 years
Response rate (complete or partial response) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Up to 2 years
Change in Akt-mediated downstream biomarkers by immunohistochemistry (IHC) | From baseline to 4 weeks at the time of surgery
  Pre-and-post treatment comparisons for correlative endpoints will be performed by the paired t-test, Wilcoxon signed-rank test, McNemar's chi-square test, or the Spearman-rank correlation coefficient, as appropriate. Exact 95% confidence intervals will be calculated to assess the precision of the obtained estimates.
Change in stem cell subpopulation | From baseline to 4 weeks at the time of surgery
  Pre-and-post treatment comparisons for correlative endpoints will be performed by the paired t-test, Wilcoxon signed-rank test, McNemar's chi-square test, or the Spearman-rank correlation coefficient, as appropriate. Exact 95% confidence intervals will be calculated to assess the precision of the obtained estimates.
Correlation between patient-specific micro-RNA signatures with response to therapy, recurrence and overall survival | At baseline and at 4 weeks at the time of surgery
  Pre-and-post treatment comparisons for correlative endpoints will be performed by the paired t-test, Wilcoxon signed-rank test, McNemar's chi-square test, or the Spearman-rank correlation coefficient, as appropriate. Exact 95% confidence intervals will be calculated to assess the precision of the obtained estimates.
Correlation of circulating melanoma endothelial cells (CECs) and circulating progenitor (CEPs) cell levels in the blood with recurrence and/or survival | Up to 2 years
  Pre-and-post treatment comparisons for correlative endpoints will be performed by the paired t-test, Wilcoxon signed-rank test, McNemar's chi-square test, or the Spearman-rank correlation coefficient, as appropriate. Exact 95% confidence intervals will be calculated to assess the precision of the obtained estimates.
Correlation between shedding of collagen cryptic epitopes with response and risk of recurrence | Up to 2 years
  Pre-and-post treatment comparisons for correlative endpoints will be performed by the paired t-test, Wilcoxon signed-rank test, McNemar's chi-square test, or the Spearman-rank correlation coefficient, as appropriate. Exact 95% confidence intervals will be calculated to assess the precision of the obtained estimates.
Pharmacokinetics of RO4929097 | At days 1 and 10
  Pre-and-post treatment comparisons for correlative endpoints will be performed by the paired t-test, Wilcoxon signed-rank test, McNemar's chi-square test, or the Spearman-rank correlation coefficient, as appropriate. Exact 95% confidence intervals will be calculated to assess the precision of the obtained estimates.
Pharmacodynamics of RO4929097 | At days 1 and 10
  Pre-and-post treatment comparisons for correlative endpoints will be performed by the paired t-test, Wilcoxon signed-rank test, McNemar's chi-square test, or the Spearman-rank correlation coefficient, as appropriate. Exact 95% confidence intervals will be calculated to assess the precision of the obtained estimates.
Impact of RO4929097 on serum markers of angiogenesis | Up to 2 years
  Pre-and-post treatment comparisons for correlative endpoints will be performed by the paired t-test, Wilcoxon signed-rank test, McNemar's chi-square test, or the Spearman-rank correlation coefficient, as appropriate. Exact 95% confidence intervals will be calculated to assess the precision of the obtained estimates.
Correlation between serum autoimmune biomarkers and clinical response | Up to 2 years
  Pre-and-post treatment comparisons for correlative endpoints will be performed by the paired t-test, Wilcoxon signed-rank test, McNemar's chi-square test, or the Spearman-rank correlation coefficient, as appropriate. Exact 95% confidence intervals will be calculated to assess the precision of the obtained estimates.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Pavlick, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - New York University Langone Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York